CLINICAL TRIAL: NCT02993523
Title: A Randomized, Double-Blind, Placebo Controlled Phase 3 Study of Venetoclax in Combination With Azacitidine Versus Azacitidine in Treatment Naïve Subjects With Acute Myeloid Leukemia Who Are Ineligible for Standard Induction Therapy
Brief Title: A Study of Venetoclax in Combination With Azacitidine Versus Azacitidine in Treatment Naïve Participants With Acute Myeloid Leukemia Who Are Ineligible for Standard Induction Therapy
Acronym: Viale-a
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-656; 2016-001466-28 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2023-01-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia; Venetoclax; Treatment Naïve; Azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 and Group 2: Placebo + Azacitidine 75 mg/m^2 (Placebo Comparator): Participants enrolled under original protocol and enrolled during or after protocol amendment 1 received venetoclax-matching placebo, orally, every day (QD), from Day 1 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, subcutaneously (SC) or intravenously (IV), QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Azacitidine; Drug: Placebo
- Group 1 and Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 (Active Comparator): Participants enrolled under original protocol and enrolled during or after protocol amendment 1 received venetoclax 100 mg, once orally, on Day 1 of Cycle 1 followed by venetoclax 200 mg, once orally, on Day 2 of Cycle 1 and venetoclax 400 mg, orally, QD, on Day 3 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, SC or IV, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Azacitidine; Drug: Venetoclax
- Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2 (Active Comparator): Participants received venetoclax 400 mg, orally, QD, from Day 1 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, SC, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Solution for subcutaneous or intravenous administration.
Drug: Venetoclax — Tablet
  Other Names: ABT-199
  Arms: Group 1 and Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2; Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2
Drug: Placebo — Matching placebo tablet
  Arms: Group 1 and Group 2: Placebo + Azacitidine 75 mg/m^2

SUMMARY:
Acute Myeloid Leukaemia (AML) is an aggressive and rare cancer of myeloid cells (a white blood cell responsible for fighting infections). Successful treatment of AML is dependent on what subtype of AML the participant has, and the age of the participant when diagnosed.

Venetoclax is an experimental drug that kills cancer cells by blocking a protein (part of a cell) that allows cancer cells to stay alive. This study is designed to see if adding venetoclax to azacitidine works better than azacitidine on its own.

This is a Phase 3, randomized, double-blind (treatment is unknown to participants and doctors), placebo controlled study in patients with AML who are >= 18 or more years old and have not been treated before. Participants who take part in this study should not be suitable for standard induction therapy (usual starting treatment). AbbVie is funding this study which will take place at approximately 180 hospitals globally and enroll approximately 400 participants.

In this study, 2/3 of participants will receive venetoclax every day with azacitidine and the remaining 1/3 will receive placebo (dummy) tablets with azacitidine.

Participants will continue to have study visits and receive treatment for as long as they are having a clinical benefit. The effect of the treatment on AML will be checked by taking blood, bone marrow, scans, measuring side effects and by completing health questionnaires. Blood and bone marrow tests will be completed to see why some people respond better than others. Additional blood tests will be completed for genetic factors and to see how long the drug remains in the body.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have confirmation of Acute Myeloid Leukemia (AML) by World Health Organization (WHO) criteria, previously untreated and be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due age or comorbidities.
* Participant must be >= 18 years of age.
* Participant must have a projected life expectancy of at least 12 weeks.
* Participant must be considered ineligible for induction therapy defined by the following:

  a. >= 75 years of age; or b. >= 18 to 74 years of age with at least one of the following comorbidities: i. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or 3; ii. Cardiac history of Congestive Heart Failure (CHF) requiring treatment or Ejection Fraction <= 50% or chronic stable angina; iii. Diffusing capacity of the Lung for Carbon Monoxide (DLCO) <= 65% or Forced Expiratory Volume in 1 second (FEV1) <= 65%; iv. Creatinine clearance >= 30 mL/min to < 45 ml/min; v. Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × Upper Limit of Normal (ULN); vi. Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy must be reviewed and approved by the AbbVie Therapeutic Medical Director during screening and before study enrollment.
* Participant must have an ECOG Performance status:

  1. 0 to 2 for Participants >= 75 years of age or
  2. 0 to 3 for Participants >= 18 to 74 years of age.
* Participant must have adequate renal function as demonstrated by a creatinine >= 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection.
* Participant must have adequate liver function as demonstrated by:

  1. aspartate aminotransferase (AST) <= 3.0 x ULN*
  2. alanine aminotransferase (ALT) <= 3.0 x ULN*
  3. bilirubin <= 1.5 x ULN* * Unless considered to be due to leukemic organ involvement

  i. Participants who are < 75 years of age may have a bilirubin of <= 3.0 x ULN
* Female participants must be either postmenopausal defined as:

  1. Age > 55 years with no menses for 12 or more months without an alternative medical cause.
  2. Age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND an follicle stimulating hormone (FSH) level >40 international units per liter (IU/L); or
  3. Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy); or
  4. Women of Childbearing Potential (WOCBP) practicing at least one protocol specified method of birth control, starting at Study Day 1 through at least 90 days after the last dose of study drug.
* Male participants who are sexually active, must agree, from Study Day 1 through at least 90 days after the last dose of study drug, to practice the protocol specified contraception. Male subjects must agree to refrain from sperm donation from initial study drug administration through at least 90 days after the last dose of study drug.
* Female participants of childbearing potential must have negative results for pregnancy test performed:

  1. At Screening with a serum sample obtained within 14 days prior to the first study drug administration, and
  2. Prior to dosing with urine sample obtained on Cycle 1 Day 1, if it has been > 7 days since obtaining the serum pregnancy test results.
* Participant must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Participant has received treatment with the following:

  1. A hypomethylating agent, venetoclax and/or chemo therapeutic agent for Myelodysplastic syndrome (MDS).
  2. Chimeric Antigen Receptor (CAR)-T cell therapy.
  3. Experimental therapies for MDS or Acute Myeloid Leukemia (AML).
  4. Current participation in another research or observational study.
* Participant has history of myeloproliferative neoplasm (MPN) including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation and AML with BCR-ABL1 translocation.
* Participant has the following:

  a. Favorable risk cytogenetics such as t(8;21), inv(16) or t(16;16) or t(15;17) as per the National Comprehensive Cancer Network (NCCN) Guidelines Version 2, 2016 for Acute Myeloid Leukemia.
* Participant has acute promyelocytic leukemia
* Participant has known active central nervous system (CNS) involvement with AML.
* Participant has known human immunodeficiency virus (HIV) infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax) HIV testing will be performed at Screening, only if required per local guidelines or institutional standards.
* Participant is known to be positive for hepatitis B or C infection [HCV Ab indicative of a previous or current infection; and/or positive HBs Ag or detected sensitivity on hepatitis B virus (HBV) deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) test for HBc Ab and/or HBs Ab positivity] with the exception of those with an undetectable viral load within 3 months screening. Hepatitis B or C testing is not required.
* Participant has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment; additional details as described in the protocol.
* Participant has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Participant has a cardiovascular disability status of New York Heart Association Class > 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
* Participant has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, any other medical condition or known hypersensitivity to any of the study medications including excipients of azacitidine that in the opinion of the investigator would adversely affect his/her participating in this study.
* Participant has a malabsorption syndrome or other condition that precludes enteral route of administration.
* Participant exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).
* Participant has a history of other malignancies within 2 years prior to study entry, with the exception of:

  1. Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  2. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  3. Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent; requires discussion with TA MD.
* Participant has a white blood cell count > 25 × 10^9/L. (Hydroxyurea or leukapheresis are permitted to meet this criterion.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2026-01-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (172):
- United States (24):
  - City of Hope /ID# 154105, Duarte, California
  - University of California, Los Angeles /ID# 154107, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center /ID# 162725, Sacramento, California
  - Emory Midtown Infectious Disease Clinic /ID# 162534, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine /ID# 201133, Chicago, Illinois
  - University of Chicago Medicine /ID# 154108, Chicago, Illinois
  - Fort Wayne Medical Oncology /ID# 157190, Fort Wayne, Indiana
  - Cotton-O'Neil Clinical Res Ctr /ID# 155136, Topeka, Kansas
  - Norton Cancer Institute /ID# 154992, Louisville, Kentucky
  - EMMC Cancer Care /ID# 154991, Brewer, Maine
  - Johns Hopkins University /ID# 154104, Baltimore, Maryland
  - Massachusetts General Hospital /ID# 200752, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 201155, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 167009, Boston, Massachusetts
  - Sepctrum Health Medical Center /ID# 159522, Grand Rapids, Michigan
  - Columbia Univ Medical Center /ID# 154101, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 165077, New York, New York
  - Duke Cancer Center /ID# 154106, Durham, North Carolina
  - University of Pittsburgh MC /ID# 154102, Pittsburgh, Pennsylvania
  - Tennessee Oncology-Nashville Centennial /ID# 200854, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center /ID# 154100, Houston, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 157191, Temple, Texas
  - University of Utah /ID# 157192, Salt Lake City, Utah
  - University Of Vermont Medical /ID# 157196, Burlington, Vermont
- Australia (7):
  - Princess Alexandra Hospital /ID# 154272, Woolloongabba, Queensland
  - Royal Adelaide Hospital /ID# 154271, Adelaide, South Australia
  - Alfred Health /ID# 154275, Melbourne, Victoria
  - St Vincent's Hospital Melbourne /ID# 155094, Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 155095, Parkville, Victoria
  - Sir Charles Gairdner Hospital /ID# 163924, Nedlands, Western Australia
  - Royal Perth Hospital /ID# 154274, Perth, Western Australia
- Austria (6):
  - Universitaetsklinikum St. Poelten /ID# 167436, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 157882, Graz, Styria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 154888, Linz, Upper Austria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 154885, Linz, Upper Austria
  - Duplicate_Landeskrankenhaus Salzburg /ID# 169719, Salzburg
  - Hanusch Krankenhaus /ID# 155676, Vienna
- Belgium (4):
  - UZ Brussel /ID# 153393, Jette, Brussels Capital
  - UCL Saint-Luc /ID# 153391, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent /ID# 153392, Ghent, Oost-Vlaanderen
  - AZ Sint-Jan Brugge /ID# 154041, Bruges
- Brazil (4):
  - Hospital de Clinicas de Porto Alegre /ID# 157779, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto - USP /ID# 153099, Ribeirão Preto, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas /ID# 157778, São Paulo, São Paulo
  - Instituto do Câncer do Estado de São Paulo - ICESP /ID# 153095, São Paulo, São Paulo
- Canada (5):
  - Tom Baker Cancer Centre /ID# 159645, Calgary, Alberta
  - St. Paul's Hospital /ID# 159644, Vancouver, British Columbia
  - Juravinski Cancer Centre /ID# 153650, Hamilton, Ontario
  - Ottawa Hospital Research Institute /ID# 153541, Ottawa, Ontario
  - Princess Margaret Cancer Centre /ID# 153651, Toronto, Ontario
- China (13):
  - Fujian Medical University Union Hospital /ID# 167314, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University /ID# 170148, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 167316, Shijiazhuang, Hebei
  - Henan Cancer Hospital /ID# 167320, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 167315, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 167493, Wuhan, Hubei
  - Jiangsu Province Hospital /ID# 167489, Nanjing, Jiangsu
  - The First Hospital of Jilin University /ID# 167490, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 167318, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 167492, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 167487, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 167317, Hangzhou, Zhejiang
  - Qilu Hospital of Shandong University /ID# 167485, Jinan
- Croatia (3):
  - Clinical Hospital Dubrava /ID# 153515, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 153383, Zagreb, City of Zagreb
  - Duplicate_Klinicki bolnicki centar Osijek /ID# 153623, Osijek, County of Osijek-Baranja
- Czechia (4):
  - Fakultni Nemocnice Brno /ID# 154019, Brno
  - Fakultni nemocnice Hradec Kralove /ID# 154021, Hradec Králové
  - Fakultni nemocnice Ostrava /ID# 154017, Ostrava
  - Fakultni nemocnice Plzen /ID# 154018, Pilsen
- Aalborg University Hospital /ID# 154047, Aalborg, North Denmark, Denmark
- Finland (3):
  - Tampere University Hospital /ID# 154963, Tampere, Pirkanmaa
  - Helsinki University Hospital /ID# 155223, Helsinki, Uusimaa
  - Turku University Hospital /ID# 154964, Turku
- France (4):
  - CHU Bordeaux - Hopital Haut Leveque /ID# 153789, Pessac, Gironde
  - Chu Angers /Id# 153792, Angers
  - AP-HP - Hopital Saint-Louis /ID# 153787, Paris
  - IUCT Oncopole /ID# 153788, Toulouse
- Germany (6):
  - Universitaetsklinikum Ulm /ID# 153054, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Frankfurt /ID# 153060, Frankfurt am Main, Hesse
  - Universitaetsklinikum Muenster /ID# 153059, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Halle (Saale) /ID# 153058, Halle
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 153056, Hamburg
  - Medizinische Hochschule Hannover /ID# 153055, Hanover
- Hungary (7):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 153812, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont /ID# 153814, Debrecen, Hajdú-Bihar
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz Josa Andras Okta /ID# 169854, Nyíregyháza, Nyiregyhaza
  - Somogy Megyei Kaposi Mor Oktato Korhaz /ID# 153813, Kaposvár, Somogy County
  - Semmelweis Egyetem /ID# 153816, Budapest
  - Duplicate_Semmelweis Egyetem /ID# 153815, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 158990, Budapest
- Israel (6):
  - The Chaim Sheba Medical Center /ID# 154173, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 154175, Tel Aviv, Tel Aviv
  - Assaf Harofeh Medical Center /ID# 158063, Be’er Ya‘aqov
  - Rambam Health Care Campus /ID# 154174, Haifa
  - Hadassah /ID# 154172, Jerusalem
  - Rabin Medical Center /ID# 154176, Petah Tikva
- Italy (10):
  - Presidio Ospedaliero Vito Fazzi /ID# 170837, Lecce, Apulia
  - Fondazione PTV Policlinico Tor Vergata /ID# 152881, Rome, Roma
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 171220, Ancona
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni /ID# 152875, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna /ID# 152883, Bologna
  - Ospedale Policlinico San Martino /ID# 158104, Genova
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 152882, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli /ID# 152879, Napoli
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli /ID# 152877, Reggio Calabria
  - Azienda Ospedaliero-Universitaria Sant'Andrea /ID# 152876, Rome
- Japan (19):
  - Aichi Cancer Center Hospital /ID# 200824, Nagoya, Aichi-ken
  - University of Fukui Hospital /ID# 167432, Yoshida-gun, Fukui
  - National Hospital Organization Kyushu Cancer Center /ID# 201111, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 169095, Fukuoka, Fukuoka
  - Gunmaken Saiseikai Maebashi Hospital /ID# 168316, Maebashi, Gunma
  - National Hospital Organization Mito Medical Center /ID# 168219, Higashi, Ibaraki
  - Hitachi General Hospital /ID# 201109, Hitachi-shi, Ibaraki
  - Duplicate_Kyoto Prefectural University of Medicine /ID# 167661, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 169259, Sendai, Miyagi
  - Nagasaki University Hospital /ID# 168632, Nagasaki, Nagasaki
  - Okayama University Hospital /ID# 204124, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital /ID# 169055, Osaka, Osaka
  - Duplicate_Kindai University Hospital /ID# 167662, Osaka-sayama-shi, Osaka
  - Saitama Medical University International Medical Center /ID# 167814, Hidaka-shi, Saitama
  - Juntendo University Hospital /ID# 168309, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital /ID# 168639, Bunkyo-ku, Tokyo
  - The Jikei University Daisan Hospital /ID# 168745, Komae-shi, Tokyo
  - NTT Medical Center Tokyo /ID# 167975, Shinagawa-ku, Tokyo
  - Yamagata University Hospital /ID# 167634, Yamagata, Yamagata
- Norway (4):
  - Akershus universitetssykehus /ID# 154279, Nordlenangen, Akershus
  - Drammen Sykehus /ID# 154280, Drammen, Buskerud
  - Haukeland University Hospital /ID# 154281, Bergen, Hordaland
  - Sykehuset Ostfold Kalnes /ID# 157755, Grålum
- Poland (3):
  - Osrodek Badan Klinicznych przy Szpitalu Specjalistycznym im. Ludwika Rydygiera w /ID# 169846, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu /ID# 153389, Wroclaw, Lower Silesian Voivodeship
  - SP ZOZ Zespol Szpitali Miejskich w Chorzowie /ID# 153385, Chorzów, Silesian Voivodeship
- Portugal (2):
  - Duplicate_Hospital de Braga /ID# 154797, Braga
  - IPO Porto FG, EPE /ID# 154138, Porto
- VA Caribbean Healthcare System /ID# 160507, San Juan, Puerto Rico
- Russia (8):
  - Kuzbass Regional Clinical Hospital /ID# 157461, Kemerovo, Kemerovo Oblast
  - Moscow State budget healthcare /ID# 155738, Moscow, Moscow
  - Nizhny Novgorod Regional Clinical Hospital named N.A. Semashko /ID# 153268, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Duplicate_Regional Oncology Dispensary /ID# 153264, Penza, Penza Oblast
  - State Institution of Health of the Ryazan Regional Clinical Hospital /ID# 157460, Ryazan, Ryazan Oblast
  - Saratov State Medical University n.a. V.I. Razumovskiy /ID# 153267, Saratov, Saratov Oblast
  - Federal State Budgetary Ins NRC for Hematology of MoH of Russian Federation /ID# 155740, Moscow
  - Samara State Medical University /ID# 157462, Samara
- South Africa (2):
  - University of Pretoria /ID# 153682, Pretoria, Gauteng
  - Albert Alberts Stem Cell Transplant Centre /ID# 153684, Pretoria, Gauteng
- South Korea (3):
  - Duplicate_Konkuk University Medical Ctr /ID# 153973, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 153675, Seoul
  - Samsung Medical Center /ID# 153674, Seoul
- Spain (8):
  - Hospital Universitario de Navarra /ID# 153254, Pamplona, Navarre
  - Hospital Clinic de Barcelona /ID# 153255, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 153193, Barcelona
  - Hospital Universitario de la Princesa /ID# 153256, Madrid
  - Hospital General Universitario Gregorio Maranon /ID# 153260, Madrid
  - Hospital Universitario 12 de Octubre /ID# 153258, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 153257, Málaga
  - Hospital Universitario y Politecnico La Fe /ID# 153259, Valencia
- Sweden (4):
  - Akademiska Sjukhuset /ID# 153034, Uppsala, Uppsala County
  - Uddevalla sjukhus /ID# 156875, Uddevalla, Västra Götaland County
  - Dup_VO Hematologi /ID# 153174, Lund
  - Karolinska University Hospital /ID# 170003, Stockholm
- Taiwan (4):
  - Changhua Christian Hospital /ID# 153899, Changhua, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 153902, Kaohsiung City
  - China Medical University Hospital /ID# 153904, Taichung
  - National Taiwan University Hospital /ID# 153900, Taipei
- Turkey (Türkiye) (3):
  - Hacettepe University Faculty of Medicine /ID# 202073, Ankara
  - Ankara Universitesi Fakultesi /ID# 155200, Ankara
  - Ondokuz Mayis Universitesi Tip /ID# 155201, Samsun
- Ukraine (4):
  - Kyiv city clinical hospital #9 /ID# 153510, Kiev, Vinnytsia Oblast
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council /ID# 153511, Dnipro
  - Kyiv Regional Onco Dispensary /ID# 153514, Kyiv
  - Poltava Reg Clin Hosp Sklifoso /ID# 153513, Poltava

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Venditti A, Hou JZ, Fenaux P, Jonas BA, Vrhovac R, Montesinos P, Garcia JS, Rizzieri D, Thirman MJ, Zhang M, Potluri J, Miller C, Dhalla M, Pullarkat V. Outcomes of patients treated with venetoclax plus azacitidine versus azacitidine alone stratified by advanced age and acute myeloid leukemia composite model. Leukemia. 2025 Nov;39(11):2697-2707. doi: 10.1038/s41375-025-02730-3. Epub 2025 Sep 5. PMID 40913104
- [Derived] Dohner H, Pratz KW, DiNardo CD, Wei AH, Jonas BA, Pullarkat VA, Thirman MJ, Recher C, Schuh AC, Babu S, Li X, Ku G, Liu Z, Sun Y, Potluri J, Dail M, Chyla B, Pollyea DA. Genetic risk stratification and outcomes among treatment-naive patients with AML treated with venetoclax and azacitidine. Blood. 2024 Nov 21;144(21):2211-2222. doi: 10.1182/blood.2024024944. PMID 39133921
- [Derived] Pollyea DA, Pratz KW, Wei AH, Pullarkat V, Jonas BA, Recher C, Babu S, Schuh AC, Dail M, Sun Y, Potluri J, Chyla B, DiNardo CD. Outcomes in Patients with Poor-Risk Cytogenetics with or without TP53 Mutations Treated with Venetoclax and Azacitidine. Clin Cancer Res. 2022 Dec 15;28(24):5272-5279. doi: 10.1158/1078-0432.CCR-22-1183. PMID 36007102
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- [Derived] Pratz KW, Chai X, Xie J, Yin L, Nie X, Montez M, Iantuono E, Downs L, Ma E. Cost-Effectiveness Analysis of Venetoclax in Combination with Azacitidine Versus Azacitidine Monotherapy in Patients with Acute Myeloid Leukemia Who are Ineligible for Intensive Chemotherapy: From a US Third Party Payer Perspective. Pharmacoeconomics. 2022 Aug;40(8):777-790. doi: 10.1007/s40273-022-01145-7. Epub 2022 Jun 13. PMID 35696071
- [Derived] Konopleva M, Thirman MJ, Pratz KW, Garcia JS, Recher C, Pullarkat V, Kantarjian HM, DiNardo CD, Dail M, Duan Y, Chyla B, Potluri J, Miller CL, Wei AH. Impact of FLT3 Mutation on Outcomes after Venetoclax and Azacitidine for Patients with Treatment-Naive Acute Myeloid Leukemia. Clin Cancer Res. 2022 Jul 1;28(13):2744-2752. doi: 10.1158/1078-0432.CCR-21-3405. PMID 35063965
- [Derived] Pollyea DA, DiNardo CD, Arellano ML, Pigneux A, Fiedler W, Konopleva M, Rizzieri DA, Smith BD, Shinagawa A, Lemoli RM, Dail M, Duan Y, Chyla B, Potluri J, Miller CL, Kantarjian HM. Impact of Venetoclax and Azacitidine in Treatment-Naive Patients with Acute Myeloid Leukemia and IDH1/2 Mutations. Clin Cancer Res. 2022 Jul 1;28(13):2753-2761. doi: 10.1158/1078-0432.CCR-21-3467. PMID 35046058
- [Derived] Pratz KW, Jonas BA, Pullarkat V, Recher C, Schuh AC, Thirman MJ, Garcia JS, DiNardo CD, Vorobyev V, Fracchiolla NS, Yeh SP, Jang JH, Ozcan M, Yamamoto K, Illes A, Zhou Y, Dail M, Chyla B, Potluri J, Dohner H. Measurable Residual Disease Response and Prognosis in Treatment-Naive Acute Myeloid Leukemia With Venetoclax and Azacitidine. J Clin Oncol. 2022 Mar 10;40(8):855-865. doi: 10.1200/JCO.21.01546. Epub 2021 Dec 15. PMID 34910556
- [Derived] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in Group 1 per original protocol stratified by age (18 - < 75, ≥ 75), and region (US, EU, Japan (JP), Rest of world (ROW)) and Group 2 during or after Amendment 1 stratified by age (18 - < 75, ≥ 75), cytogenetic risk (intermediate, poor) and region (US, EU, China, JP, ROW).
Pre-assignment Details: Total of 443 participants were enrolled. 433 participants were randomized in Group 1 and Group 2 to receive placebo or venetoclax 100/200/400mg+azacitidine 75mg/m^2. 10 participants in open-label China cohort received venetoclax 400 mg + azacitidine 75 mg/m^2 up to data cut-off date: 01 December 2021. This study is ongoing.
Groups:
- Group 1: Placebo + Azacitidine 75 mg/m^2: Participants enrolled under original protocol received venetoclax-matching placebo, orally, once daily (QD), from Day 1 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, subcutaneously (SC) or intravenously (IV), QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
- Group 1: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2: Participants enrolled under original protocol received venetoclax 100 mg, once orally, on Day 1 of Cycle 1 followed by venetoclax 200 mg, once orally, on Day 2 of Cycle 1 and venetoclax 400 mg, orally, QD, on Day 3 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, SC or IV, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
- Group 2: Placebo + Azacitidine 75 mg/m^2: Participants received venetoclax-matching placebo, orally, QD, from Day 1 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, SC or IV, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
- Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2: Participants received venetoclax 100 mg, once orally, on Day 1 of Cycle 1 followed by venetoclax 200 mg, once orally, on Day 2 of Cycle 1 and venetoclax 400 mg, orally, QD, from Day 3 to Day 28 of each 28-day cycle along with azacitidine 75 mg/m^2, SC or IV, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
Period: Overall Study
Arm/Group | Group 1: Placebo + Azacitidine 75 mg/m^2 | Group 1: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 | Group 2: Placebo + Azacitidine 75 mg/m^2 | Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 | Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2
Started | 1 | 1 | 145 | 286 | 10
Completed | 0 | 0 | 1 | 48 | 4
Not Completed | 1 | 1 | 144 | 238 | 6
Not completed — Withdrew Consent | 0 | 0 | 2 | 9 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 6 | 0
Not completed — Death | 1 | 1 | 138 | 222 | 6
Not completed — Reason not Specified | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all Group 1 and 2 participants randomized by Interactive Voice Response System (IVRS)/Interactive Web Response System (IWRS) (exclude the open-label China safety cohort). Open-Label China Safety Cohort included participants who received at least one dose of venetoclax.
Groups:
- Group 1: Placebo + Azacitidine 75 mg/m^2: Participants enrolled under original protocol received venetoclax-matching placebo, orally, QD, from Day 1 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, SC or IV, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
- Total: Total of all reporting groups
Arm/Group | Group 1: Placebo + Azacitidine 75 mg/m^2 | Group 1: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 | Group 2: Placebo + Azacitidine 75 mg/m^2 | Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 | Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2 | Total
Number analyzed (Participants) | 1 | 1 | 145 | 286 | 10 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (NA) — Standard deviation (SD) was not estimable for 1 participant. | 65.0 (NA) — SD was not estimable for 1 participant. | 75.1 (5.70) | 75.6 (6.08) | 70.2 (7.44) | 75.2 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 58 | 114 | 4 | 177
  Male | 0 | 1 | 87 | 172 | 6 | 266
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 33 | 66 | 10 | 109
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3 | 0 | 6
  White | 0 | 1 | 109 | 217 | 0 | 327
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the number of days from the date of randomization to the date of death. Log rank test was used to compare the OS distribution between two treatment arms. Cox regression was used to report the hazard ratio.
Time Frame: From the study start up to death or alive or lost to follow-up (up to approximately 4.8 years; data cut off date: 1 December 2021)
Population: Full Analysis Set included all Group 2 participants randomized by IVRS/IWRS (exclude the open-label China safety cohort).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2: Placebo + Azacitidine 75 mg/m^2 | Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 145 | 286
months | 9.6 [7.4 to 12.7] | 14.7 [12.1 to 18.7]
Statistical Analysis 1: Comparison: Group 2: Placebo + Azacitidine 75 mg/m^2 vs Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2; Test type: Superiority; p < 0.001, Log Rank — Stratified log-rank test stratified by age (18 - < 75, ≥ 75) and cytogenetic risk (intermediate, poor); Hazard Ratio (HR) = 0.580, 95% CI 2-sided [0.465 to 0.723] — HR from Cox proportional hazards model stratified by age (18 - < 75, ≥ 75) and cytogenetic risk (intermediate, poor)

2. Primary Outcome: Percentage of Participants With Complete Remission (CR) and Complete Remission With Incomplete Marrow Recovery (CRi)
Description: CR and CRi was calculated based on current International Working Group (IWG) criteria. CR is defined as absolute neutrophil count >10^3/ microliter (mcL), platelets >10^5/mcL, red cell transfusion independence, and bone marrow with <5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of ≤10^3/mcL or platelets ≤10^5/mcL. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: From the study start up to death (up to approximately 4.8 years; data cut-off date: 1 December 2021)
Population: Full Analysis Set included all Group 2 participants randomized by IVRS/IWRS (exclude the open-label China safety cohort). Open-Label China Safety Cohort included participants who received at least one dose of venetoclax. Data is reported for Group 2 and Open-label China Cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: Placebo + Azacitidine 75 mg/m^2 | Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 | Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2
Number analyzed (Participants) | 145 | 286 | 10
percentage of participants
  CR | 17.9 [12.1 to 25.2] | 38.8 [33.1 to 44.7] | 60.0 [26.2 to 87.8]
  CRi | 11.0 [6.4 to 17.3] | 28.0 [22.8 to 33.6] | 20.0 [2.5 to 55.6]
Statistical Analysis 1: Comparison: Group 2: Placebo + Azacitidine 75 mg/m^2 vs Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test stratified by age (18 - < 75, ≥ 75) and cytogenetic risk (intermediate, poor)

3. Secondary Outcome: Event-free Survival (EFS)
Description: EFS will be defined as the number of days from randomization to the date of progressive disease, relapse from CR or CRi, treatment failure or death from any cause.
Time Frame: Measured up to 2 years after the last participant is randomized
Reporting Status: Not Posted, anticipated posting 2027-01

4. Secondary Outcome: Global Health Status/Quality of Life (GHS/QoL)
Description: Improvement in GHS/QoL will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) and European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core (EORTC QLQ-C30).
Time Frame: Measured at participant's Day 1 of Cycle 1 (each cycle is 28 days) and at Day 1 of every Cycle thereafter for up to 2 years following the last subject last visit
Reporting Status: Not Posted, anticipated posting 2027-01

5. Secondary Outcome: Percentage of Participants Achieving Composite Complete Remission (CR or CRi)
Description: This will be calculated based on current International Working Group (IWG) criteria. CR is defined as absolute neutrophil count > 10^3/mcL, platelets > 10^5/mcL, red cell transfusion independence, and bone marrow with < 5% blasts. CRi is defined as bone marrow with less than 5% blasts, and absolute neutrophils of <= 10^3/mcL or platelets <= 10^5/mcL.
Time Frame: Up to 6 months after the first 225 participants are randomized
Reporting Status: Not Posted, anticipated posting 2027-01

6. Secondary Outcome: Complete Remission or Complete Remission With Partial Hematologic Recovery Rate (CR+CRh)
Description: A response of CRh is defined as Bone marrow with <5% blasts, peripheral blood neutrophil count >0.5*10^3/mcL and peripheral blood platelet count >0.5*10^5/mcL.
Time Frame: Measured up to 2 years after the last participant is randomized
Reporting Status: Not Posted, anticipated posting 2027-01

7. Secondary Outcome: Post Baseline Transfusion Independence Rate
Description: Transfusion Independence is defined as a period of 56 days with no transfusion between first dose of study drug and the last dose of study drug + 30 days. The rate of conversion for red blood cells (RBC) and platelets is defined as percentage of participants being post-baseline transfusion independent from baseline transfusion dependence.
Time Frame: Measured up to 2 years after the last participant is randomized
Reporting Status: Not Posted, anticipated posting 2027-01

8. Secondary Outcome: Complete Remission (CR) Rate
Description: The percentage of participants with complete remission (CR) will be calculated based on the modified IWG criteria for AML.
Time Frame: Measured up to 2 years after the last participant is randomized
Reporting Status: Not Posted, anticipated posting 2027-01

9. Secondary Outcome: Fatigue/Quality of Life (QoL)
Description: Fatigue QoL will be assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) Cancer Fatigue Short Form (SF) 7a global fatigue score
Time Frame: Measured at participant's Day 1 of Cycle 1 (each cycle is 28 days) and at Day 1 of every Cycle thereafter for up to 2 years following the last participant last visit
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Time Frame: From the study start until data cut-off date: 01 December 2021 (up to approximately 4.8 years)
Description: Safety analysis set included all Group 1 and Group 2 participants (exclude the open-label China safety cohort) who took at least one dose of venetoclax/placebo and azacitidine combination. As pre-specified in SAP the data is reported combined for both Group 1 and Group 2 participants who received either placebo plus azacitidine or venetoclax plus azacitidine. Open-Label China Safety Cohort included participants who received at least one dose of venetoclax in combination with azacitidine.
Groups:
- Group 1 and Group 2: Placebo + Azacitidine 75 mg/m^2: Participants enrolled under original protocol and enrolled during or after protocol amendment 1 received venetoclax-matching placebo, orally, QD, from Day 1 to Day 28 of each 28 day cycle along with azacitidine 75 mg/m^2, SC or IV, QD for 7 days from Day 1 of each 28-day cycle until documented disease progression, unacceptable toxicity, withdrawal of consent, or other protocol criteria for discontinuation (whichever occurred first).
Arm/Group | Group 1 and Group 2: Placebo + Azacitidine 75 mg/m^2 | Group 1 and Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 | Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 140/144 | 226/283 | 6/10
Serious Adverse Events (participants affected / at risk) | 111/144 | 242/283 | 7/10
Other Adverse Events (participants affected / at risk) | 137/144 | 279/283 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 and Group 2: Placebo + Azacitidine 75 mg/m^2 (N=144) | Group 1 and Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 (N=283) | Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2 (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 9 (13) | 19 (23) | 0 (0)
CYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 15 (21) | 88 (132) | 2 (2)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4) | 14 (15) | 3 (3)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 14 (14) | 3 (4)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (4) | 2 (2) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 13 (15) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 3 (3) | 7 (8) | 1 (1)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
MYOCARDIAL OEDEMA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
TORSADE DE POINTES (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (4) | 6 (6) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
GASTRODUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERTROPHIC ANAL PAPILLA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
NECROTISING COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PALATAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PROCTITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 4 (4) | 0 (0)
CATHETER SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 2 (2) | 4 (4) | 0 (0)
DISCOMFORT (General disorders) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 5 (6) | 5 (6) | 0 (0)
IMPAIRED SELF-CARE (General disorders) | 0 (0) | 1 (1) | 0 (0)
INCARCERATED HERNIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 2 (2) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (2) | 2 (3) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 9 (10) | 0 (0)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
SUDDEN DEATH (General disorders) | 0 (0) | 2 (2) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 (2) | 3 (4) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CONGESTION (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATITIS CHOLESTATIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
ABSCESS FUNGAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACINETOBACTER BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ALVEOLAR OSTEITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 3 (5) | 0 (0)
ANORECTAL CELLULITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
ASPERGILLUS INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 7 (9) | 0 (0)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
BRONCHITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS MORAXELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
BURKHOLDERIA INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CANDIDA SEPSIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
CANDIDURIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 4 (4) | 7 (9) | 0 (0)
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS ORBITAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CITROBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CORONA VIRUS INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
DERMATITIS INFECTED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 6 (9) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROBACTER PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 7 (8) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 2 (2) | 9 (10) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FUNGAL SEPSIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
GINGIVITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTIOUS THYROIDITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 2 (2) | 8 (9) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 3 (3) | 10 (10) | 2 (2)
MEDICAL DEVICE SITE CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PAROTITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PERICORONITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PHARYNGOTONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 35 (46) | 55 (71) | 0 (0)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PROTEUS INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
PSOAS ABSCESS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
PULMONARY MYCOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PULMONARY NOCARDIOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PULPITIS DENTAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RECTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 12 (14) | 20 (29) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 8 (11) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
SYSTEMIC CANDIDA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC MYCOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (6) | 10 (11) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
WATERHOUSE-FRIDERICHSEN SYNDROME (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ARTERIAL BYPASS OCCLUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 3 (4) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
INCISION SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (2) | 2 (2) | 0 (0)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 2 (2) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 3 (3) | 0 (0)
CLOSTRIDIUM TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
COMPUTERISED TOMOGRAM HEAD ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 2 (3) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 3 (3) | 0 (0)
POLYOMAVIRUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCUS TEST POSITIVE (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
SERONEGATIVE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SOFT TISSUE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
ERYTHROLEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2) | 0 (0)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 3 (4) | 0 (0)
COMA (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0)
MOTOR NEURONE DISEASE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 6 (6) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 5 (5) | 5 (5) | 0 (0)
AZOTAEMIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0)
RENAL MASS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
STRANGURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX SPONTANEOUS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIAL HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
COELIAC ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHAGIC VASCULITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 2 (3) | 5 (5) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 and Group 2: Placebo + Azacitidine 75 mg/m^2 (N=144) | Group 1 and Group 2: Venetoclax 100 mg/200 mg/400 mg + Azacitidine 75 mg/m^2 (N=283) | Open Label China Cohort: Venetoclax 400 mg + Azacitidine 75 mg/m^2 (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 24 (30) | 68 (102) | 6 (11)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 12 (16) | 33 (44) | 3 (3)
LEUKOPENIA (Blood and lymphatic system disorders) | 20 (46) | 54 (133) | 10 (20)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (6) | 8 (16) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 38 (66) | 107 (245) | 5 (6)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 57 (94) | 120 (246) | 6 (15)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 13 (15) | 22 (26) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 5 (5) | 1 (1)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 8 (8) | 1 (1)
CONJUNCTIVAL DISORDER (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
KERATITIS (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
OPTIC ATROPHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 3 (4) | 1 (1)
XEROPHTHALMIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 (4) | 6 (8) | 2 (3)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 (7) | 9 (11) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 (14) | 34 (42) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (6) | 17 (19) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 55 (66) | 121 (158) | 7 (9)
DIARRHOEA (Gastrointestinal disorders) | 46 (65) | 122 (182) | 5 (5)
DYSPEPSIA (Gastrointestinal disorders) | 7 (7) | 20 (23) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 3 (3) | 5 (6) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 3 (4) | 6 (6) | 2 (2)
GINGIVAL SWELLING (Gastrointestinal disorders) | 1 (2) | 2 (2) | 2 (2)
HAEMORRHOIDS (Gastrointestinal disorders) | 6 (6) | 29 (31) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 53 (65) | 123 (178) | 4 (6)
STOMATITIS (Gastrointestinal disorders) | 9 (10) | 32 (39) | 0 (0)
VOMITING (Gastrointestinal disorders) | 33 (44) | 84 (128) | 5 (9)
ASTHENIA (General disorders) | 12 (17) | 45 (55) | 0 (0)
FATIGUE (General disorders) | 24 (29) | 61 (83) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 10 (11) | 17 (19) | 1 (1)
INJECTION SITE REACTION (General disorders) | 11 (14) | 13 (24) | 4 (5)
INJECTION SITE SWELLING (General disorders) | 1 (1) | 0 (0) | 1 (1)
MALAISE (General disorders) | 2 (2) | 15 (21) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 26 (30) | 70 (96) | 0 (0)
PAIN (General disorders) | 4 (6) | 16 (20) | 0 (0)
PYREXIA (General disorders) | 30 (43) | 66 (93) | 2 (5)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 3 (4) | 9 (15) | 1 (2)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
ANAL INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
GASTROINTESTINAL FUNGAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
GINGIVITIS (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1) | 11 (11) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 5 (8) | 17 (21) | 0 (0)
ORAL HERPES (Infections and infestations) | 7 (7) | 17 (18) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 8 (8) | 19 (19) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
TINEA INFECTION (Infections and infestations) | 1 (2) | 2 (3) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 (15) | 25 (29) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 7 (9) | 22 (34) | 1 (2)
BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 12 (13) | 16 (22) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 8 (10) | 33 (54) | 0 (0)
ADENOSINE DEAMINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11 (15) | 24 (34) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 12 (16) | 22 (31) | 3 (4)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (5) | 15 (25) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 5 (6) | 21 (28) | 4 (6)
BLOOD CREATININE INCREASED (Investigations) | 8 (13) | 13 (15) | 2 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 2 (2) | 7 (8) | 4 (7)
C-REACTIVE PROTEIN INCREASED (Investigations) | 4 (4) | 16 (17) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (3) | 7 (11) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2) | 7 (12) | 1 (2)
PLATELET COUNT DECREASED (Investigations) | 3 (9) | 13 (24) | 1 (1)
WEIGHT DECREASED (Investigations) | 18 (22) | 42 (61) | 4 (5)
DECREASED APPETITE (Metabolism and nutrition disorders) | 26 (29) | 78 (101) | 6 (7)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 (7) | 12 (14) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 15 (16) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 (2) | 9 (10) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 7 (8) | 8 (9) | 4 (5)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 13 (15) | 23 (31) | 2 (5)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 9 (10) | 19 (27) | 5 (6)
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 43 (59) | 84 (125) | 8 (13)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5 (7) | 24 (28) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 6 (6) | 16 (20) | 2 (2)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 17 (23) | 36 (46) | 2 (2)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (7) | 35 (43) | 3 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (9) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 (14) | 25 (32) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 18 (19) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 15 (19) | 23 (27) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 11 (14) | 37 (51) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 11 (13) | 1 (1)
HEADACHE (Nervous system disorders) | 12 (13) | 34 (38) | 1 (2)
PARAESTHESIA (Nervous system disorders) | 2 (2) | 8 (10) | 1 (1)
POOR QUALITY SLEEP (Nervous system disorders) | 4 (5) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 15 (17) | 36 (39) | 3 (4)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 8 (10) | 21 (27) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 36 (40) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 37 (49) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 24 (30) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 28 (38) | 1 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 27 (29) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 17 (20) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (6) | 15 (17) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 8 (8) | 18 (19) | 0 (0)
PRURIGO (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (7) | 28 (34) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 9 (9) | 31 (40) | 3 (3)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4) | 24 (27) | 0 (0)
AORTIC ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMATOMA (Vascular disorders) | 9 (14) | 16 (21) | 0 (0)
HYPERTENSION (Vascular disorders) | 12 (14) | 30 (32) | 2 (3)
HYPOTENSION (Vascular disorders) | 7 (9) | 23 (31) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT02993523/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT02993523/SAP_001.pdf